CLINICAL TRIAL: NCT05056441
Title: ENTYVIO® Real-World Outcomes in Bio-naïve Crohn's Disease Patients in Belgium, Australia, and Switzerland: An EVOLVE Observational Expansion Study
Brief Title: A Study of Real-World Outcomes of People With Crohn's Disease (CD)
Acronym: EVOLVE
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Vedolizumab-5066
Record Dates: First submitted 2021-08-27; First posted 2021-09-24 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Crohn Disease
Keywords: Drug Therapy
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Vedolizumab: Biologic-naïve participants diagnosed with CD, who have initiated vedolizumab treatment will be observed from the data of diagnosis of CD until the date of index when vedolizumab treatment was initiated during the eligibility period until the earliest of chart abstraction initiation, death or last contact with the site. Index date is defined as the date when vedolizumab treatment was initiated.
- Cohort 2: Ustekinumab: Biologic-naïve participants diagnosed with CD, who have initiated ustekinumab treatment will be observed from the data of diagnosis of CD until the date of index when ustekinumab treatment was initiated during the eligibility period until the earliest of chart abstraction initiation, death or last contact with the site. Index date is defined as the date when ustekinumab treatment was initiated.

SUMMARY:
The main aim of this study is to compare long-term remission in participants receiving vedolizumab (VDZ) and those receiving ustekinumab (UST).

In this study, the study doctors will review each participant's past medical records. This study is about collecting existing information only; participants will not receive treatment or need to visit a study doctor during this study.

DETAILED DESCRIPTION:
This is a non-interventional, retrospective study of participants with CD. The study will review the medical charts of participants who have initiated the treatment with vedolizumab and ustekinumab or another biologic agent (post- index).

The study will aim to enroll approximately 700 participants, with 350 participants in each of the following cohorts:

* Cohort 1: Vedolizumab
* Cohort 2: Ustekinumab

The data for participants will be collected in two main periods:

* Pre-Index Event Period: From the date of diagnosis of CD until the date of index when vedolizumab or ustekinumab was initiated during the eligibility period.
* Post-Index Event Period: From one day post-index when vedolizumab or ustekinumab was initiated during the eligibility period until chart abstraction initiation, unless the date of death or loss to follow-up is before the date of chart abstraction initiation.

This multi-center study will be conducted in Belgium, Australia, and Switzerland. The overall time for data collection in the study will be approximately 12 months and the long-term duration of the study is approximately 36 months.

ELIGIBILITY:
Inclusion Criteria:

1. Has a diagnosis of CD documented in the medical records.
2. Has received at least one dose of vedolizumab or ustekinumab at one of the participating study sites during the eligibility period.
3. Was biologic-naïve (no prior biologic use for any pathology, including CD) at the time of index event.
4. Has completed induction phase and has a minimum of a six-month duration between the date of the index event and the date of chart abstraction initiation and was still under active care at the site six months post-index date.

Exclusion Criteria:

1. Has received vedolizumab or ustekinumab as part of a clinical trial in their lifetime (includes index event).
2. Has initiated index treatment as combination therapy with two biologic agents.
3. Has received previous treatment with biologic agents for CD or conditions other than CD ever in their lifetime.
4. Has medical chart empty or missing.
5. Part or all of the participant's index treatment was received at a different site, and the participant's medical chart pertaining to this care is not accessible.
6. Has received a subcutaneous formulation of ustekinumab for induction (that is, a subcutaneous induction dose of ustekinumab prior to ustekinumab's approval for CD in the study countries).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Biologic-naïve CD participants who initiated biologic treatment with vedolizumab or ustekinumab (index event) during the eligibility period.
Sampling Method: Non-Probability Sample
Enrollment: 623 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Cumulative Rates of Clinical Remission Over 36 Months Compared Between VDZ and UST Cohorts | Baseline up to 36 months post-index date
  Clinical remission will be defined as Crohn's Disease Activity Index (CDAI) score less than (<) 150 points, or if unknown, Harvey-Bradshaw Index (HBI) Overall score less than or equal to (<=) 4 points, or if unknown, Modified HBI (mHBI) score <=4 points, or if unknown, changes in biomarker assessments (C-reactive Protein, Fecal Calprotectin, and albumin) or remission status recorded in medical chart as 'in remission'. CDAI score <150 indicates quiescent disease and >450 indicates extremely severe disease. HBI consisted of 5 clinical parameters: general well-being, abdominal pain, number of liquid stools per day, abdominal mass, and complications. mHBI consisted of 4 clinical parameters- general well-being, abdominal pain, number of liquid stools per day and additional manifestation. HBI and mHBI total score will be sum of individual parameters, score ranges 0 to no pre-specified maximum score as it depends on number of liquid stools, where higher scores is more severe disease.

SECONDARY OUTCOMES:
Cumulative Rates of Clinical Response Over 36 Months Compared Between VDZ and UST Cohorts | Baseline up to 36 months post-index date
  Clinical response will be defined as CDAI positive change in score from baseline, or if unknown, HBI overall score decrease of >=3 points from baseline, or if unknown, Modified HBI score decrease of >=3 points from baseline, or if unknown, changes in biomarker assessments (CRP, FCP, and albumin) or treatment response recorded in the medical chart as 'complete response' or 'partial response'. CDAI score <150 indicates quiescent disease and >450 indicates extremely severe disease. HBI consisted of 5 clinical parameters: general well-being, abdominal pain, number of liquid stools per day, abdominal mass, and complications. mHBI consisted of 4 clinical parameters- general well-being, abdominal pain, number of liquid stools per day and additional manifestation. HBI and mHBI total score will be sum of individual parameters, score ranges 0 to no pre-specified maximum score as it depends on number of liquid stools, where higher scores is more severe disease.
Cumulative Rates of Clinical Remission Over 30 Months Compared Between VDZ and UST Cohorts | Baseline up to 30 months post-index date
  Clinical remission will be defined as CDAI score <150 points, or if unknown, HBI Overall score of <=4 points, or if unknown, mHBI score of <=4 points, or if unknown, changes in biomarker assessments (CRP, FCP, and albumin) or remission status recorded in the medical chart as 'in remission'. CDAI score <150 indicates quiescent disease and >450 indicates extremely severe disease. HBI consisted of 5 clinical parameters: general well-being, abdominal pain, number of liquid stools per day, abdominal mass, and complications. mHBI consisted of 4 clinical parameters- general well-being, abdominal pain, number of liquid stools per day and additional manifestation. HBI and mHBI total score will be sum of individual parameters, score ranges 0 to no pre-specified maximum score as it depends on number of liquid stools, where higher scores is more severe disease.
Cumulative Rates of Mucosal Healing Over 36 Months Compared Between VDZ and UST Cohorts | Baseline up to 36 months post-index date
  Mucosal healing will be defined as endoscopic assessment score = 0 or 1 (that is, normal or inactive disease or mild disease), or if unknown, Simple Endoscopic Score for Crohn's Disease [SES-CD] score of <3, 'lack of ulceration' defined by one or more of the following endoscopic procedure findings either selection of 'no ulcers' or free-text indication of 'lack of ulceration', or if unknown, one or more endoscopic procedure findings indicating inactive disease (no findings/no active disease, no erosion, no ulcers, no inflammation or inflammatory activity, or no pathological findings), with higher scores indicating more severe disease. The score for each endoscopic variable is sum of values obtained for each segment. The SES-CD total is sum of the 4 endoscopic variable scores from 0 to 56, where higher scores indicate more severe disease.
Cumulative Rates of Deep Remission Over 36 Months Compared Between VDZ and UST Cohorts | Baseline up to 36 months post-index date
  Deep remission (clinical remission and mucosal healing) is defined as CDAI score <150 and SES-CD score <3. CDAI is scoring system for the assessment of CD activity, index values of 150 and below are associated with quiescent disease; values above that indicate active disease and values above 450 are seen with extremely severe disease. The SES-CD evaluates 4 endoscopic variables (ulcer size, percentage of the surface area affected, and stenosis in 5 colonic segments evaluated during ileocolonoscopy (ileum, right colon, transverse colon, left colon, and rectum). The SES-CD total is the sum of the 4 endoscopic variable scores from 0 to 56, where higher scores indicate more severe disease.
Cumulative Rates of Corticosteroid (CS)-free Remission Over 36 Months Compared Between VDZ and UST Cohorts | Baseline up to 36 months post-index date
  CS-free remission is defined as participants using oral corticosteroids at baseline who have discontinued corticosteroids and have clinical remission up to 36-months.
Cumulative Rates of CS-free Response Over 36 Months Compared Between VDZ and UST Cohorts | Baseline up to 36 months post-index date
  Corticosteroid-free response is defined as participants using oral corticosteroids at baseline who have discontinued oral corticosteroids and have clinical response up to 36-months.
Time to Treatment Switching Compared Between VDZ and UST Cohorts | From index event up to a maximum of 36 months post-index date
  Time to Treatment Switching is defined as time from index treatment initiation until a participant initiates subsequent treatments.
Time to Treatment Discontinuation Compared Between VDZ and UST Cohorts | From index event up to a maximum of 36 months post-index date
  Time to Treatment Discontinuation is defined as time from index treatment initiation until participant discontinues index treatment without switching to subsequent treatments.
Time to Dose Escalation Compared Between VDZ and UST Cohorts | From index event up to a maximum of 36 months post-index date
  Time to Dose Escalation is defined as time from index treatment initiation until increase in index treatment frequency or dose and/or treatment frequency for >=2 consecutive drug administrations.
Incidence Rate of Adverse Events (AEs) Compared Between VDZ and UST Cohorts | From the index event (Baseline) to the earliest date of chart abstraction initiation, death or last contact with the site (up to approximately Month 6 post-index date)
  Incidence rate of AE will be measured in per 100 person-years. 100 person-years will be used as it is a method that can account for large among-participant variations in follow-up time.
Incidence Rate of Serious Adverse Events (SAEs) Compared Between VDZ and UST Cohorts | From the index event (Baseline) to the earliest date of chart abstraction initiation, death or last contact with the site (up to approximately Month 6 post-index date)
  Incidence rate of SAEs will be measured in per 100 person-years. 100 person-years will be used as it is a method that can account for large among-participant variations in follow-up time. SAE is defined as an AE that either results in death, was a life threatening event), requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, results in a congenital anomaly/birth defect, or is a medically important event in the opinion of the physician.
Incidence Rate of Serious Infections (SIs) Compared Between VDZ and UST Cohorts | From the index event (Baseline) to the earliest date of chart abstraction initiation, death or last contact with the site (up to approximately Month 6 post-index date)
  Incidence rate of SIs will be measured in per 100 person-years. 100 person-years will be used as it is a method that can account for large among-participant variations in follow-up time. SI is defined as an SAE that is an infection.
Incidence Rate of Emergency Department (ED) Visits Compared Between VDZ and UST Cohorts | From the index event (Baseline) to the earliest date of chart abstraction initiation, death or last contact with the site (up to approximately Month 12 post-index date)
  Incidence rate of ED will be measured in per 100 person-years. 100 person-years will be used as it is a method that can account for large among-participant variations in follow-up time.
Incidence Rate of CD-related Hospitalizations Compared Between VDZ and UST Cohorts | From the index event (Baseline) to the earliest date of chart abstraction initiation, death or last contact with the site (up to approximately Month 12 post-index date)
  Incidence rate of CD-related hospitalizations will be measured in per 100 person-years. 100 person-years will be used as it is a method that can account for large among-participant variations in follow-up time. and CD-related Hospitalizations is defined as hospitalization with reason for hospitalization related to CD.
Incidence Rate of CD-related Surgical Procedures compared between VDZ and UST cohorts | From the index event (Baseline) to the earliest date of chart abstraction initiation, death or last contact with the site (up to approximately Month 12 post-index date)
  Incidence rate of CD-related surgical procedures will be measured in per 100 person-years. 100 person-years will be used as it is a method that can account for large among-participant variations in follow-up time. CD-related surgical procedures are defined as types of surgeries that are related to CD.
Incidence Rate of Disease Exacerbations Compared Between VDZ and UST Cohorts | From the date of initiation of subsequent line treatment up to the earliest date of chart abstraction initiation, death or last contact with the site (up to a maximum of 36 months post-index date)
  Incidence rate of disease exacerbations will be measured in per 100 person-years. 100 person-years will be used as it is a method that can account for large among-participant variations in follow-up time. Exacerbations are defined as disease flares documented in the participant's medical chart.
Time to Treatment Switching of Subsequent Line Treatments Compared Between VDZ and UST Cohorts | From the date of initiation of subsequent line treatment up to the earliest date of chart abstraction initiation, death or last contact with the site (up to a maximum of 36 months post-index date)
  Subsequent line treatment is defined as biologic and advanced therapy regimen(s) for participants who discontinued biologic vedolizumab or ustekinumab and initiated one or more biologic and advanced therapies, post-index treatment discontinuation.
Time to Treatment Discontinuation of Subsequent Line Treatments Compared Between VDZ and UST Cohorts | From the date of initiation of subsequent line treatment up to the earliest date of chart abstraction initiation, death or last contact with the site (up to a maximum of 36 months post-index date)
  Subsequent line treatment is defined as biologic and advanced therapy regimen(s) for participants who discontinued biologic vedolizumab or ustekinumab and initiated one or more biologic and advanced therapies, post-index treatment discontinuation.
Time to Dose Escalation of Subsequent Line Treatments Compared Between VDZ and UST Cohorts | From the date of initiation of subsequent line treatment up to the earliest date of chart abstraction initiation, death or last contact with the site (up to a maximum of 36 months post-index date)
  Subsequent line treatment is defined as biologic and advanced therapy regimen(s) for participants who discontinued biologic vedolizumab or ustekinumab and initiated one or more biologic and advanced therapies, post-index treatment discontinuation.
Cumulative Rates of Clinical Response of Subsequent Line Treatments Compared Between VDZ and UST Cohorts | From the date of initiation of subsequent line treatment up to the earliest date of chart abstraction initiation, death or last contact with the site (up to a maximum of 36 months post-index date)
  Clinical response defined as CDAI positive change in score from baseline, if unknown, HBI overall score decrease >=3 points from baseline, if unknown, mHBI score decrease >=3 points from baseline, if unknown, changes in CRP, FCP, albumin or treatment response as complete response/partial response. CDAI score <150 indicates quiescent disease, >450 indicates extremely severe disease. HBI includes general well-being, abdominal pain, number of liquid stools per day, abdominal mass, complications. mHBI includes general well-being, abdominal pain, number of liquid stools/day, additional manifestation. HBI and mHBI total score is sum of individual parameters, score ranges 0 to no pre-specified maximum score, as it depends on number of liquid stools, higher scores means severe disease. Subsequent line treatment: biologic and advanced therapy regimen for participants who discontinued biologic VDZ and UST, initiated 1 or more biologic, advanced therapies, post-index treatment discontinuation.
Cumulative Rates of Clinical Remission of Subsequent Line Treatments Compared Between VDZ and UST Cohorts | From the date of initiation of subsequent line treatment up to the earliest date of chart abstraction initiation, death or last contact with the site (up to a maximum of 36 months post-index date)
  Clinical remission defined as CDAI score <150 points, or if unknown, HBI Overall score of <=4 points, or if unknown, mHBI score of <=4 points, or if unknown, changes in CRP, FCP, and albumin or remission status recorded in the medical chart as 'in remission'. CDAI score <150 indicates quiescent disease and >450 indicates extremely severe disease. HBI includes: general well-being, abdominal pain, number of liquid stools/day, abdominal mass, complications. mHBI includes- general well-being, abdominal pain, number of liquid stools/day and additional manifestation. HBI and mHBI total score will be sum of individual parameters, score ranges 0 to no pre-specified maximum score as it depends on number of liquid stools, where higher scores is more severe disease. Subsequent line treatment is defined as biologic and advanced therapy regimen(s) for participants who discontinued biologic VDZ or UST and initiated one or more biologic and advanced therapies, post-index treatment discontinuation.
Cumulative Rates of Mucosal Healing of Subsequent Line Treatments Compared Between VDZ and UST Cohorts | From the date of initiation of subsequent line treatment up to the earliest date of chart abstraction initiation, death or last contact with the site (up to a maximum of 36 months post-index date)
  Mucosal healing defined as endoscopic score = 0 or 1 (normal or inactive disease or mild disease), or if unknown, Simple Endoscopic Score for Crohn's Disease [SES-CD] score of <3, 'lack of ulceration' defined by one or more of following endoscopic procedure findings either selection of 'no ulcers' or free-text indication of 'lack of ulceration', or if unknown, one or more endoscopic procedure findings: inactive disease (no findings/no active disease, no erosion, no ulcers, no inflammation or inflammatory activity, or no pathological findings), higher scores more severe disease. Score for each endoscopic variable is sum of values obtained for each segment. SES-CD total is sum endoscopic variable scores: 0 to 56, higher scores indicate more severe disease. Subsequent line treatment is defined as biologic and advanced therapy regimen(s) for participants who discontinued biologic VDZ or UST and initiated one or more biologic and advanced therapies, post-index treatment discontinuation.
Cumulative Rates of Deep Remission of Subsequent Line Treatments Compared Between VDZ and UST Cohorts | From the date of initiation of subsequent line treatment up to the earliest date of chart abstraction initiation, death or last contact with the site (up to a maximum of 36 months post-index date)
  Deep remission (clinical remission and mucosal healing) is defined as CDAI score <150 and SES-CD score <3. CDAI is scoring system for the assessment of CD activity, index values of 150 and below are associated with quiescent disease; values above that indicate active disease and values above 450 are seen with extremely severe disease. The SES-CD evaluates 4 endoscopic variables (ulcer size, percentage of the surface area affected, and stenosis in 5 colonic segments evaluated during ileocolonoscopy (ileum, right colon, transverse colon, left colon, and rectum). The SES-CD total is the sum of the 4 endoscopic variable scores from 0 to 56, where higher scores indicate more severe disease. Subsequent line treatment is defined as biologic and advanced therapy regimen(s) for participants who discontinued biologic vedolizumab or ustekinumab and initiated one or more biologic and advanced therapies, post-index treatment discontinuation.
Cumulative Rates of Corticosteroid (CS)-free Remission of Subsequent Line Treatments Compared Between VDZ and UST Cohorts | From the date of initiation of subsequent line treatment up to the earliest date of chart abstraction initiation, death or last contact with the site (up to a maximum of 36 months post-index date)
  CS-free remission is defined as participants using oral corticosteroids at baseline. Subsequent line treatment is defined as biologic and advanced therapy regimen(s) for participants who discontinued biologic vedolizumab or ustekinumab and initiated one or more biologic and advanced therapies, post-index treatment discontinuation.
Cumulative Rates of CS-free Response of Subsequent Line Treatments Compared Between VDZ and UST Cohorts | From the date of initiation of subsequent line treatment up to the earliest date of chart abstraction initiation, death or last contact with the site (up to a maximum of 36 months post-index date)
  Corticosteroid-free response is defined as participants using oral corticosteroids at baseline. Subsequent line treatment is defined as biologic and advanced therapy regimen(s) for participants who discontinued biologic vedolizumab or ustekinumab and initiated one or more biologic and advanced therapies, post-index treatment discontinuation.
Incidence Rate of AEs of Subsequent Line Treatments Compared Between VDZ and UST Cohorts | From the date of initiation of subsequent line treatment up to the earliest date of chart abstraction initiation, death or last contact with the site (up to a maximum of 36 months post-index date)
  Incidence rate of AE will be measured in per 100 person-years. 100 person-years will be used as it is a method that can account for large among-participant variations in follow-up time. Subsequent line treatment is defined as biologic and advanced therapy regimen(s) for participants who discontinued biologic vedolizumab or ustekinumab and initiated one or more biologic and advanced therapies, post-index treatment discontinuation.
Incidence Rate of SAEs of Subsequent Line Treatments Compared Between VDZ and UST Cohorts | From the date of initiation of subsequent line treatment up to the earliest date of chart abstraction initiation, death or last contact with the site (up to a maximum of 36 months post-index date)
  Incidence rate of SAEs will be measured in per 100 person-years. 100 person-years will be used as it is a method that can account for large among-participant variations in follow-up time. SAE is defined as an AE that either results in death, was a life threatening event), requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, results in a congenital anomaly/birth defect, or is a medically important event in the opinion of the physician. Subsequent line treatment is defined as biologic and advanced therapy regimen(s) for participants who discontinued biologic vedolizumab or ustekinumab and initiated one or more biologic and advanced therapies, post-index treatment discontinuation.
Incidence Rate of SIs of Subsequent Line Treatments Compared Between VDZ and UST Cohorts | From the date of initiation of subsequent line treatment up to the earliest date of chart abstraction initiation, death or last contact with the site (up to a maximum of 36 months post-index date)
  Incidence rate of SIs will be measured in per 100 person-years. 100 person-years will be used as it is a method that can account for large among-participant variations in follow-up time. SI is defined as an SAE that is an infection. Subsequent line treatment is defined as biologic and advanced therapy regimen(s) for participants who discontinued biologic vedolizumab or ustekinumab and initiated one or more biologic and advanced therapies, post-index treatment discontinuation.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (31):
- Australia (13):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - John Hunter Hospital, New Lambton, New South Wales
  - Royal Brisbane & Women's Hospital, Herston, Queensland
  - Mater Misericordiae Health Services, South Brisbane, Queensland
  - Integrated Gut Health Pty Ltd, Taringa, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - Monash Health, Monash Medical Centre, Clayton, Victoria
  - Royal Melbourne Hospital, East Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - St John of God Hospital Subiaco, Subiaco, Western Australia
- Belgium (13):
  - Imelda VZW, Bonheiden, Antwerpen
  - UZ Antwerpen, Edegem, Antwerpen
  - Hopital Erasme, Anderlecht, Brussels Capital
  - Centre Hospitalier Universitaire Ambroise Pare, Mons, Hainaut
  - CHWAPI Tournai, Tournai, Hainaut
  - AZ Sint-Lucas, Ghent, Oost-Vlaanderen
  - UZ Gent, Ghent, Oost-Vlaanderen
  - UZ Leuven, Leuven, Vlaams Brabant
  - AZ Groeninge, Kortrijk, West-Vlaanderen
  - AZ Delta, Roeselare, West-Vlaanderen
  - CHU St-Pierre, Brussels
  - Centre Hospitalier Chretien MontLegia, Liège
  - CHU de Liege, Liège
- Switzerland (5):
  - Clarunis Bauchzenturm, Basel, Basel-Stadt (de)
  - Inselspital Bern, Bern, Bern (de)
  - Intesto KLG Gastroenterologische Praxis Crohn-Colitis-Zentrum, Bern, Bern (de)
  - Stadtspital Triemli Zurich, Zurich, Zurich (de)
  - Universitatsspital Zurich, Zurich, Zurich (de)

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Christensen B, Scharl M, Bressler B, Khan Z, Halchenko Y, Gisler C, Kamble P, Adsul S, Farhat Z, Ferrante M. Real-World Clinical Effectiveness and Safety of Vedolizumab and Ustekinumab in Biologic-Naive Patients With Early or Late Crohn's Disease: Results From the EVOLVE Expansion Study. Crohns Colitis 360. 2025 Jul 9;7(3):otaf031. doi: 10.1093/crocol/otaf031. eCollection 2025 Jul. PMID 40641824
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/614e34bbc15195002c0ba31b